CLINICAL TRIAL: NCT04650880
Title: A Randomized Double-blind Controlled Trial on the Effect of Vitamin D on Ovulation Rate of Women With Polycystic Ovary Syndrome
Brief Title: Effect of Vitamin D on Ovulation Rate in Women With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwong Wah Hospital (Other); Princess Margaret Hospital, Hong Kong (Other Government); Pamela Youde Nethersole Eastern Hospital (Other); The Queen Elizabeth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW20-004
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome; Anovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D 50,000 IU/ week for 4 weeks, followed by 50,000 IU once every 2 weeks for 52 weeks Those who remain anovulatory after 6 months will be treated with a 6-month course of letrozole (2.5mg to 7.5mg for 5 days per cycle titrated according to response) for ovulation induction.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo tablets with same external appearance for 52 weeks Those who remain anovulatory after 6 months will be treated with a 6-month course of letrozole (2.5mg to 7.5mg for 5 days per cycle titrated according to response) for ovulation induction.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D supplementation
  Arms: Vitamin D
Other: Placebo — Placebo tablets with the same external appearance
  Arms: Placebo

SUMMARY:
This is a randomized double-blind controlled trial on the effect of vitamin D supplementation to assess the ovulation rate of women with polycystic ovary syndrome (PCOS) and other reproductive, endocrine and metabolic outcomes after one year of treatment.

DETAILED DESCRIPTION:
The hypothesis is that vitamin D supplementation results in significant improvement in the ovulation rate of women with PCOS either spontaneously or with oral ovulation induction agent.

Anovulatory women with PCOS diagnosed by the Rotterdam criteria will be recruited.

Participants will be randomized to the (1) vitamin D group or (2) placebo group. Those in the vitamin D group will take vitamin D 50,000 IU/ week for 4 weeks, followed by 50,000IU once every 2 weeks for 52 weeks, whereas those in the placebo group will take placebo tablets with the same external appearance. Those who remain anovulatory after 6 months will be treated with a 6-month course of letrozole (2.5mg to 7.5mg for 5 days per cycle titrated according to response) for ovulation induction.

The primary outcome is the ovulation rate and will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* Aged 18-40 years
* Irregular long menstrual cycles (>35 days)
* PCOS according to the Rotterdam criteria
* Agree for transvaginal ultrasound

Exclusion Criteria:

* Use of hormonal medication (including contraception) within 3 months prior to study inclusion, except the use of a progestogen to induce withdrawal bleeding every 3 months
* History of any medical condition or medications that may predispose to vitamin D sensitivity, altered vitamin D metabolism and/ or hypercalcemia, including active tuberculosis or current therapy for tuberculosis, sarcoidosis, history of renal/ ureteral stones, parathyroid disease, renal or liver failure or current use of anti-convulsants
* Use of insulin-sensitizing drugs, lipid lowering drugs or anti-hypertensive
* Anticipated to use the above medications in the coming one year
* Known type 2 diabetes mellitus
* Refusal to join the study
* Abnormal blood calcium level

For those on supplements, we asked them to stop their own supplements.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ovulation rate | 12 months
  Serum progesterone

SECONDARY OUTCOMES:
Change in serum 25(OH)D level | 12 months
  Serum 25(OH)D
Pregnancy rate | 12 months
  Positive urine or serum hCG test
Live birth rate | 12 months
  Delivery of a baby after 22 completed weeks of gestational age, or with birth weight of 500 grams if the gestation age is unknown, which shows evidence of life
Change in serum anti-Mullerian hormone level | 12 months
  serum AMH level
Change in antral follicle count | 12 months
  Antral follicle count measured by transvaginal/ transrectal ultrasound
Androgen indices | 12 months
  serum androgen and androstenedione levels, SHBG
Body mass index | 12 months
  Height in cm, weight in kg, to calculate the body mass index (kg/m^2)
Change in waist and hip circumference | 12 months
  waist and hip circumference in cm
Rate of diabetes mellitus/ impaired glucose intolerance | 12 months
  Measured by fasting and 2 hour glucose (post 75g OGTT)
Change in systolic and diastolic blood pressure | 12 months
  Blood pressure

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Kwong Wah Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Time Frame: starting 6 months after publication
Access Criteria: review by investigators

REFERENCES:
- [Derived] Ko JKY, Yung SSF, Lai SF, Wan RSF, Wong CKY, Wong K, Cheung CL, Ng EHY, Li RHW. Effect of vitamin D in addition to letrozole on the ovulation rate of women with polycystic ovary syndrome: protocol of a multicentre randomised double-blind controlled trial. BMJ Open. 2024 Apr 29;14(4):e070801. doi: 10.1136/bmjopen-2022-070801. PMID 38684265